CLINICAL TRIAL: NCT00996346
Title: Phase I/II Study of Irinotecan and Temsirolimus in Patients With Refractory Sarcomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Original PI left institution and sponsor decided to end support.
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0909; 3066K1 (Other: Wyeth); 3066K1-1208 (Other: Wyeth); 20091334 (Other: Western IRB); NCI-2011-01940 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Sarcoma
Keywords: INST 0909; Irinotecan; Temsirolimus; refractory sarcomas; 3066K1; 3066K1-1208; 20091334
MeSH Terms: conditions — Sarcoma | interventions — Irinotecan; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Irinotecan&Temsirolimus:Arm 1, Level 1 (Experimental): Arm 1, Level 1: Irinotecan intravenously at 80 mg/m2 + Temsirolimus intravenously at 15 mg on a weekly basis for 3 consecutive doses followed by one week of rest.
  One cycle is four weeks.
  Interventions: Drug: Irinotecan&Temsirolimus:Arm1, Level 1
- Irinotecan&Temsirolimus:Arm 1, Level 2 (Experimental): Arm 1, Level 2: Irinotecan intravenously at 80 mg/m2 + Temsirolimus intravenously at 20 mg on a weekly basis for 3 consecutive doses followed by one week of rest.
  One cycle is four weeks.
  Interventions: Drug: Irinotecan&Temsirolimus:Arm 1, Level 2
- Irinotecan&Temsirolimus:Arm 2, Level 1 (Experimental): Arm 1, Level 2: Irinotecan intravenously at 50 mg/m2 + Temsirolimus intravenously at 25 mg on a weekly basis for 3 consecutive doses followed by one week of rest.
  One cycle is four weeks.
  Interventions: Drug: Irinotecan&Temsirolimus:Arm 2, Level 1

INTERVENTIONS:
Drug: Irinotecan&Temsirolimus:Arm1, Level 1 — Irinotecan is given first over 60 minutes followed by temsirolimus over 30 minutes. No intrapatient dose escalations are allowed. Treatment continues until disease progression or intolerable side effects develop.
  Other Names: Irinotecan = Camptosar, Campto, or CPT-11; Temsirolimus = Toricel or CCI-779
  Arms: Irinotecan&Temsirolimus:Arm 1, Level 1
Drug: Irinotecan&Temsirolimus:Arm 1, Level 2 — Irinotecan is given first over 60 minutes followed by temsirolimus over 30 minutes. No intrapatient dose escalations are allowed. Treatment continues until disease progression or intolerable side effects develop.
  Other Names: Irinotecan = Camptosar, Campto, or CPT-11; Temsirolimus = Toricel or CCI-779
  Arms: Irinotecan&Temsirolimus:Arm 1, Level 2
Drug: Irinotecan&Temsirolimus:Arm 2, Level 1 — Irinotecan is given first over 60 minutes followed by temsirolimus over 30 minutes. No intrapatient dose escalations are allowed. Treatment continues until disease progression or intolerable side effects develop.
  Other Names: Irinotecan = Camptosar, Campto, or CPT-11; Temsirolimus = Toricel or CCI-779
  Arms: Irinotecan&Temsirolimus:Arm 2, Level 1

SUMMARY:
Refractory soft tissue sarcoma remains a difficult malignancy to treat. The mammalian target of rapamycin (mTOR) is an enzyme that plays an important role in cancer cell survival. mTOR inhibitors, like temsirolimus, have shown activity in sarcoma. Irinotecan is a chemotherapy drug that has also been used to treat sarcoma. However, it is unknown whether combining these two drugs would result in improved efficacy with acceptable toxicity.

Therefore, the goal of this phase I study is to determine the maximum tolerated dose (MTD) and toxicity profile of combination temsirolimus and irinotecan both administered intravenously on a weekly basis to refractory soft tissue sarcoma patients.

DETAILED DESCRIPTION:
Mammalian target of rapamycin (mTOR) inhibitors are anti-neoplastic agents with a wide potential range of clinical applications. The topoisomerase I inhibitor irinotecan is a potent DNA damaging drug. mTOR appears to enhance cancer cell survival following DNA damage, so it's reasonable to expect that mTOR inhibition combined with irinotecan may result in synergistic activity.

This is a single arm, non-randomized phase I trial of temsirolimus (an mTOR inhibitor) and irinotecan (a topoisomerase I inhibitor) in refractory soft tissue sarcoma patients. Successive groups of three patients will be entered at escalating dose levels. Irinotecan and temsirolimus will be administered weekly for three weeks followed by one week of rest. One course will therefore be four weeks. No intra-patient dose escalation will be allowed. Each patient will be treated until disease progression or intolerable side effects develop. Dose limiting toxicities will be assessed and the maximum tolerated dose will be reported.

Note that this trial was originally designed as a phase I/II study, but only the phase I portion was completed and will be reported.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 10 years of age or older with biopsy proven advanced soft tissue sarcoma, who have failed at least one prior treatment for metastatic disease are eligible if there is measurable or evaluable disease per Response Evaluation Criteria In Solid Tumors (RECIST).
* Patients must have a life expectancy of at least 12 weeks.
* Prior surgery or radiotherapy for primary tumor is acceptable but must be completed at least 4 weeks from study entry, and patient should have completely recovered from such procedures.
* Patients must have a Zubrod performance status of 0-2.
* Patients (or their legal guardian) must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of ≥ 1500 cells/mm3, hemoglobin > 8 g/dl, platelet count ≥ 100 000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have a normal hepatic function with a total bilirubin < the upper limit of normal and Serum glutamic oxaloacetic transaminase (SGOT) or Serum glutamic pyruvic transaminase (SGPT) < 2 times the upper limit of normal, and adequate renal function as defined by a serum creatinine ≤ 1.5 upper limit of normal.
* Fasting total cholesterol level < 350 mg/dL and triglyceride level < 400 mg/dL is required.
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and at least for 3 months.

Patients with brain metastases are eligible if they have been appropriately treated,are asymptomatic and no longer require corticosteroids.

Exclusion Criteria:

* Pregnant women or nursing mothers are not eligible.
* Patients must not receive any other concurrent chemotherapy or radiation during this trial.
* Patients with severe medical illnesses such as uncontrolled diabetes, active infections, or uncontrolled psychiatric illnesses are not eligible.
* Patients with known hypersensitivity to temsirolimus or sirolimus, receiving concomitant antitumor therapy, or anticonvulsant therapy, or cardiac antiarrhythmic drugs are not eligible.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monte Shaheen, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Result] Verschraegen CF, Movva S, Ji Y, Schmit B, Quinn RH, Liem B, Bocklage T, Shaheen M. A phase I study of the combination of temsirolimus with irinotecan for metastatic sarcoma. Cancers (Basel). 2013 Apr 11;5(2):418-29. doi: 10.3390/cancers5020418. PMID 24216984
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org
- See also: University of New Mexico Cancer Center — http://cancer.unm.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between October, 2009, and May, 2011
Groups:
- Irinotecan&Temsirolimus:Arm 2, Level 1: Arm 1, Level 2: Irinotecan intravenously at 50 mg/m2 + Temsirolimus intravenously at 25 mg on a weekly basis for 3 consecutive doses followed by one week of rest.
Period: Overall Study
Arm/Group | Irinotecan&Temsirolimus:Arm 1, Level 1 | Irinotecan&Temsirolimus:Arm 1, Level 2 | Irinotecan&Temsirolimus:Arm 2, Level 1
Started | 6 | 8 | 3
Completed | 6 | 8 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irinotecan&Temsirolimus:Arm 1, Level 1 | Irinotecan&Temsirolimus:Arm 1, Level 2 | Irinotecan&Temsirolimus:Arm 2, Level 1 | Total
Number analyzed (Participants) | 6 | 8 | 3 | 17
Age, Continuous [Median (Full Range); unit: years] | 60.5 [48 to 69] | 47.5 [25 to 72] | 56 [56 to 64] | 56 [25 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 1 | 8
  Male | 3 | 4 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Irinotecan
Description: The MTD is the dose preceding that at which at least 2 out of 3 patients in the treatment group experience a dose limiting toxicity (DLT). DLT is defined as grade 3 neutropenia on retreatment day, a grade 4 febrile neutropenia, a drug-related grade 3 or 4 non-hematologic toxicity (except fatigue, nausea, vomiting or grade 3 hypersensitivity reaction) or a grade 2 or greater motor or sensory neuropathy
Time Frame: Up to 1 month
Measure: Number; unit: milligrams/meter squared
Groups:
- Irinotecan&Temsirolimus:All Arms: Data from the dose escalation in all three arms is used to calculate the maximum tolerated dose (MTD).
  In all three arms, Irinotecan and temsirolimus will be repeated weekly x 3 doses followed by one week of rest. One course will be four weeks.
  The treatment consists of:
  Irinotecan at 50 - 80 mg/m2 weekly, for three weeks + Temsirolimus at 15 - 25 mg weekly, for three weeks.
  The specific doses of Irinotecan are 50, 65, or 80 mg/m2 The specific doses of Temsirolimus are 15, 20, or 25 mg
Arm/Group | Irinotecan&Temsirolimus:All Arms
Number analyzed (Participants) | 17
milligrams/meter squared | 80

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Temsirolimus
Description: as for outcome 1
Time Frame: Up to 1 month
Measure: Number; unit: milligrams
Arm/Group | Irinotecan&Temsirolimus:All Arms
Number analyzed (Participants) | 17
milligrams | 20

ADVERSE EVENTS:
Arm/Group | Irinotecan&Temsirolimus:Arm 1, Level 1 | Irinotecan&Temsirolimus:Arm 1, Level 2 | Irinotecan&Temsirolimus:Arm 2, Level 1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan&Temsirolimus:Arm 1, Level 1 (N=6) | Irinotecan&Temsirolimus:Arm 1, Level 2 (N=8) | Irinotecan&Temsirolimus:Arm 2, Level 1 (N=3)
Allergic reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Runny nose) (General disorders) | 3 (3) | 1 (1) | 0 (0)
Hemoglobin levels decreased (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 0 (0)
Hemolysis (red blood cell destruction) (Blood and lymphatic system disorders) | 0 (0) | 4 (6) | 0 (0)
Leukocytes decreased (Blood and lymphatic system disorders) | 1 (1) | 6 (16) | 2 (2)
Lymphocytes decreased (Blood and lymphatic system disorders) | 0 (0) | 8 (22) | 2 (2)
Neutrophils decreased (Blood and lymphatic system disorders) | 2 (3) | 2 (10) | 2 (2)
Platelets decreased (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (5) | 3 (4) | 2 (2)
Fever (General disorders) | 2 (2) | 1 (1) | 0 (0)
Weight loss (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatology/Skin - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Itching) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4)
Anorexia (Loss of appetite) (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (4) | 2 (4)
Hemorrhage nasal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Muscle inflammation) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Throat Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Edema: limbs (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 3 (5) | 0 (0)
Hypercalcemia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Investigations) | 2 (4) | 6 (7) | 2 (2)
Hypoalbuminemia (Investigations) | 0 (0) | 4 (6) | 1 (1)
Hypocalcemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Investigations) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesemia (Investigations) | 0 (0) | 3 (4) | 0 (0)
Hyponatremia (Investigations) | 0 (0) | 4 (4) | 0 (0)
Hypophosphatemia (Investigations) | 0 (0) | 1 (2) | 0 (0)
INR (Prothrombin time) (Investigations) | 1 (3) | 1 (2) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 3 (4) | 0 (0)
Prothromboplastin time (Investigations) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Extraocular muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gait abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3)
Headache (General disorders) | 1 (2) | 3 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (2) | 1 (1) | 1 (2)
Ear, nose and throat examination abnormal (General disorders) | 1 (1) | 1 (2) | 0 (0)
Abdominal pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Joint pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (General disorders) | 1 (1) | 3 (9) | 0 (0)
Bone pain (General disorders) | 0 (0) | 1 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Thrombosis (Vascular disorders) | 1 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No